CLINICAL TRIAL: NCT02198300
Title: Regular Drug Eluting Stent Versus Dedicated Bifurcation Sirolimus-eluting Stent BiOSS LIM in Coronary Bifurcation Treatment - Randomized POLBOS II Study.
Brief Title: DES Versus BiOSS LIM - POLBOS II Study
Acronym: POLBOS II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Jacek Bil, MD, PhD, Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.1
Record Dates: First submitted 2014-07-20; First posted 2014-07-23 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease
Keywords: dedicated bifurcation stent; sirolimus eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon; Biosensing Techniques; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rDES Group (Active Comparator): regular drug-eluting stent implantation in coronary lesion within bifurcation LucChopin Xience Promus Resolute Integrity Biomatrix Prolim
  Interventions: Procedure: Coronary angioplasty with stent implantation; Drug: Dual antipletlet therapy (DAPT)
- BiOSS LIM Group (Experimental): BiOSS LIM® stent implantation into coronary lesion within bifurcation.
  Interventions: Procedure: Coronary angioplasty with stent implantation; Drug: Dual antipletlet therapy (DAPT)

INTERVENTIONS:
Procedure: Coronary angioplasty with stent implantation
  Other Names: device: LucChopin (Balton, Poland); device: Xience (Abbot Vascular); device: Promus (Boston Scientific); device: Resolute Integrity (Medtronic); device: Biomatrix (Biosensors); device: Prolim (Balton, Poland)
Drug: Dual antipletlet therapy (DAPT) — DAPT given to each patient before stent implantation
  Other Names: acetysalicylic acid; clopidogrel

SUMMARY:
Coronary bifurcation lesions pose therapeutic problems during percutaneous coronary interventions (PCI) and are associated with higher rates of periprocedural complications as well as higher rates of in-stent restenosis and stent thrombosis. Provisional T-stenting (PTS) is the best treatment strategy at the moment. However, the optimal approach to coronary bifurcations treatment is still a subject of debate, especially when the side branch is large, not easily accessible and narrowed by a long lesion. One of the proposed alternatives are dedicated bifurcation stents (DBS). However, there is large scarcity of randomized trials with DBS. POLBOS II study is continuation of POLBOS I (POLish Bifurcation Optimal Stenting) study, in which paclitaxel-eluting stent BiOSS Expert® (Balton, Poland) was assessed. Now performance of sirolimus-eluting stent BiOSS LIM® (Balton, Poland) is verified.

DETAILED DESCRIPTION:
After signing the informed consent patients were randomly assigned to one of two treatment strategies: BiOSS LIM® stent implantation or rDES implantation (envelope randomization, 1:1). If the patient was enrolled to rDES Group there was a second randomization: with or without final kissing ballooning (FKB). Clinical follow-up was performed with office visits or telephone contacts at 1 and 12 months after intervention. Adverse events were monitored throughout the study period. Follow-up coronary angiography was performed at 12 months unless clinically indicated earlier.

ELIGIBILITY:
Inclusion Criteria:

* stable coronary artery disease (CAD) or non-ST-segment elevation acute coronary syndrome (NSTE-ACS)
* age ≥ 18 years old,
* de novo coronary bifurcation lesion (including unprotected LMS),
* MV diameter ≥ 2.5 mm and SB diameter ≥ 2.0 mm assessed by visual estimation.

Exclusion Criteria:

* ST-elevation myocardial infarction (STEMI),
* bifurcations with Medina type 0,0,1,
* serum creatinine level ≥ 2.0 mg/dl,
* inability to take dual antiplatelet therapy for 12 months,
* left ejection fraction ≤ 30%
* lack of an informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
MACE | 12 months
  Cumulative rate of major adverse cardiovascular events (MACE) including cardiac death, myocardial infarction (MI) and repeated revascularization of the target lesion (TLR)

SECONDARY OUTCOMES:
cardiac death | 12 months
all-cause death | 12 months
MI | 12 months
  myocardial infarction
TLR | 12 months
  target lesion revascularization
TVR | 12 months
  target vessel revascularization
LLL | 12 months
  late lumen loss

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Gil, MD, PhD, Principal Investigator — Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Locations (1):
- Central Clinical Hospital of the Ministry of Interior, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Background] Bil J, Gil RJ, Vassilev D, Rzezak J, Kulawik T, Pawlowski T. Dedicated bifurcation paclitaxel-eluting stent BiOSS Expert(R) in the treatment of distal left main stem stenosis. J Interv Cardiol. 2014 Jun;27(3):242-51. doi: 10.1111/joic.12119. Epub 2014 Apr 7. PMID 24708143
- [Background] Vassilev D, Mateev H, Alexandrov A, Stankev M, Rigatelli G, Gil RJ. Stenting below-the-knee bifurcations with dedicated bifurcation stent BiOSS Lim - first in man case report. Cardiovasc Revasc Med. 2014 Apr;15(3):171-7. doi: 10.1016/j.carrev.2013.09.005. Epub 2013 Oct 22. PMID 24157310
- [Background] Gil RJ, Bil J, Michalek A, Vassiliev D, Costa RA. Comparative analysis of lumen enlargement mechanisms achieved with the bifurcation dedicated BiOSS) stent versus classical coronary stent implantations by means of provisional side branch stenting strategy: an intravascular ultrasound study. Int J Cardiovasc Imaging. 2013 Dec;29(8):1667-76. doi: 10.1007/s10554-013-0264-0. Epub 2013 Jul 19. PMID 23868287
- [Background] Gil RJ, Vassilev D, Michalek A, Kern A, Formuszewicz R, Dobrzycki S, Wojcik J, Lesiak M, Kardaszewicz P, Lekston A. Dedicated paclitaxel-eluting bifurcation stent BiOSS(R) (bifurcation optimisation stent system): 12-month results from a prospective registry of consecutive all-comers population. EuroIntervention. 2012 Jul 20;8(3):316-24. doi: 10.4244/EIJV8I3A50. PMID 22829507
- [Background] Vassilev D, Gil R, Milewski K. Bifurcation Optimisation Stent System (BiOSS Lim) with sirolimus elution: results from porcine coronary artery model. EuroIntervention. 2011 Sep;7(5):614-20. doi: 10.4244/EIJV7I5A98. PMID 21930466
- [Derived] Gil RJ, Kern A, Formuszewicz R, Inigo Garcia LA, Dobrzycki S, Vassilev D, Bil J. 6-year results of BiOSS stents in coronary bifurcation treatment. Eur J Clin Invest. 2021 Aug;51(8):e13555. doi: 10.1111/eci.13555. Epub 2021 Mar 29. PMID 33782985